CLINICAL TRIAL: NCT07298603
Title: Nutrition Intervention in PCOS: Clinical, Biochemical, and Symptomatic Effects of Different Dietary Models
Brief Title: Nutrition Intervention for Women With Polycystic Ovary Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Menşure Nur ÇELİK, Principal Investigator, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2ODM.0.20.08/569
Record Dates: First submitted 2025-11-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: PCOS- Polycystic Ovary Syndrome; Nutrition Intervention; Nutrition Assessment
Keywords: polycystic ovary syndrome; FertilOMed Diet; Mediterranean Diet; dietary intervention; reproductive health; Quality of life; oxidative stress
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean Diet group (Active Comparator): Participants follow Mediterranean Diet
  Interventions: Other: MedDiet
- FertilOMed Diet (Experimental): Participants follow Fertility-Optimized Mediterranean Diet
  Interventions: Other: FertilOMed Diet
- Control (No Intervention): Participants receive standard dietary recommendations

INTERVENTIONS:
Other: FertilOMed Diet — FertilOMed Diet (Experimental): Participants will follow the FertilOMed Diet, which is based on the standard Mediterranean Diet guidelines, with required consumption of specific foods and adherence to recommended food group portions. Dietary adherence will be monitored through food diaries and follow-up consultations.
  Arms: FertilOMed Diet
Other: MedDiet — Mediterranean Diet (Active Comparator): Participants will follow a standard Mediterranean Diet for the duration of the study. Dietary adherence will be monitored through food diaries and follow-up consultations.
  Arms: Mediterranean Diet group

SUMMARY:
The goal of this clinical trial is to evaluate whether different dietary models can improve clinical, metabolic, hormonal, anthropometric, and quality-of-life parameters in women with polycystic ovary syndrome (PCOS).

The main questions it aims to answer are:

* Do the Mediterranean Diet and the FertilOMed Diet (Fertility-Optimized Mediterranean Diet) lead to significant improvements in these parameters compared to the control group?
* Does the FertilOMed Diet lead to greater improvements compared to the standard Mediterranean Diet? Study Description: This randomized controlled intervention study will be conducted between November 2025 and March 2026 at the Samsun Training and Research Hospital, Department of Obstetrics and Gynecology, Women's Health Outpatient Clinics. Necessary institutional permissions have been obtained for conducting the study at these sites.

Participants: Women diagnosed with PCOS who meet the inclusion criteria and volunteer to participate will be included in the study.

Interventions:

Participants will be randomly assigned to one of the following groups:

* Mediterranean Diet group
* FertilOMed Diet group (Fertility-Optimized Mediterranean Diet)
* Control group (standard dietary recommendations) Researchers will compare these groups to determine whether the dietary interventions improve clinical, biochemical, and symptomatic outcomes in women with PCOS.

DETAILED DESCRIPTION:
This study will include volunteer female individuals who have applied to the Gynecology and Obstetrics outpatient clinic of the Gynecology and Obstetrics Department of Samsun Training and Research Hospital, diagnosed with PCOS by a physician, and selected according to inclusion and exclusion criteria. Women who meet the criteria will be informed about the study's objectives and methodology, and those who agree to participate will be asked to sign a consent form. Individuals will be assigned to control and intervention groups, matched by age and BMI. Care will be taken to ensure that the groups are matched by age and body mass index (BMI). At the beginning of the study, a questionnaire containing sociodemographic information, general health information, dietary habits, physical activity status, sleep habits, morningness-eveningness scale, PCOS-50 Quality of Life scale, Beck depression scale, SF-36 scale, and food consumption record will be administered to the individuals via face-to-face interviews by the researcher. Initial anthropometric measurements of the female volunteers will be taken by the researcher using appropriate techniques. Additionally, biochemical findings will be obtained from hospital records at the beginning and end of the study. Volunteers, matched by age and BMI, were included in the control and intervention groups and will be followed for 12 weeks. Individuals in the control group will receive only medical treatment throughout the study period. They will be free to make food choices without energy restrictions (ad libitum). No dietary intervention will be implemented. Individuals in the intervention groups will receive ad libitum nutrition education and brochures about the diet's content, in addition to their medical treatment. Individuals in both intervention groups will not be restricted in their daily dietary energy intake.

During the 12-week follow-up period, individuals will be closely monitored through mobile applications and routine follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with PCOS according to the Rotterdam Criteria, between the ages of 20 and 45,
* Having a Body Mass Index (BMI) of 18.50-35.00 kg/m2,
* Not having used antibiotics and/or probiotics in the last month,
* Signing a voluntary consent form.

Exclusion Criteria:

* Being younger than 20 years old or older than 45 years old with PCOS diagnosis,
* Having a BMI of ≤18.50 kg/m2 and ≥35.00 kg/m2,
* Being pregnant or breastfeeding,
* Using alcohol,
* Having used antibiotics and/or probiotics in the last month,
* Having had bariatric surgery,
* Having type 1 diabetes, type 2 diabetes, Cushing's syndrome, hypothyroidism, androgen tumors, active cancer, or a gastrointestinal system or malabsorption disease,
* Having used hormonal contraceptives or insulin sensitivity-enhancing medications within 3 months before the study start,
* Having used antioxidant supplements such as vitamin C within 1 month before the study start,
* Having a Mediterranean Diet Adherence Score (MEDAS) of ≥10,
* Those who did not give their consent after reading the informed consent form.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Hormonal Profile | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  The primary outcome measure of this study is to evaluate holistic changes in the reproductive-metabolic profile of individuals with PCOS following the dietary intervention. This composite outcome includes coordinated changes in hormonal balance (e.g., FSH, LH, Estradiol, Progesterone, 17-Hydroxyprogesterone, DHEAS, T4, TSH, Prolactin, SHBG, AMH, Total Testosterone, and FAI). All parameters will be measured at baseline and after the 12-week dietary intervention, and changes will be analyzed to determine the overall impact of the applied dietary model. These parameters will be obtained by scanning the participants' routine results from their file information.
Changes in Metabolic Profile | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  The primary outcome measure of this study is to evaluate holistic changes in the reproductive-metabolic profile of individuals with PCOS following the dietary intervention. This composite outcome includes coordinated changes in metabolic profile (e.g., , AST, ALT, Hemogram, D Vitamini, B12 Vitamini, SHBG, HbA1c, AMH, Total Testosteron, Glukoz, İnsülin, HOMA IR, HDL, LDL, Trigliserit, Total Kolesterol). All parameters will be measured at baseline and after the 12-week dietary intervention, and changes will be analyzed to determine the overall impact of the applied dietary model. These parameters will be obtained by scanning the participants' routine results from their file information.
Changes in Oxidative Stress | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  The primary outcome measure of this study is to evaluate holistic changes in the reproductive-metabolic profile of individuals with PCOS following the dietary intervention. This composite outcome includes coordinated changes in hormonal balance (e.g.,TAC, Vit C, SOD, Catalase, Glutathione Peroxidase (GPx) and Malondialdehyde (MDA)). All parameters will be measured at baseline and after the 12-week dietary intervention, and changes will be analyzed to determine the overall impact of the applied dietary model. These parameters will be determined by performing validated commercial ELISA kits in accordance with the manufacturer's instructions and evaluating with a microplate reader.

SECONDARY OUTCOMES:
Changes in Body Mass Index (BMI) | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Body mass index (BMI) will be calculated using weight (kg) and height (m²). Although weight and height will be measured, only BMI (kg/m²) will be reported as the outcome variable. Changes in BMI from baseline to the end of the 12-week dietary intervention will be evaluated to assess the impact of the intervention on anthropometric status.
Change in Waist Circumference | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Anthropometric parameter used to assess central adiposity.
Change in Hip Circumference | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Anthropometric parameter used to evaluate lower-body fat distribution.
Change in Waist-to-Hip Ratio | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Derived anthropometric index reflecting fat distribution.
Change in Neck Circumference | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Anthropometric indicator associated with upper-body fat distribution.
Change in Body Fat Percentage | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Body fat percentage will be measured using the TANITA BC-545N bioelectrical impedance device under standardized conditions (8-hour fasting, light clothing, removal of metal/electronic items). Changes from baseline to Week 12 will be assessed.
Change in Lean Mass | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Lean mass will be measured using the TANITA BC-545N device under standardized measurement conditions. Changes from baseline to Week 12 will be evaluated.
Change in Muscle Mass | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Muscle mass will be assessed via TANITA BC-545N using standardized fasting and measurement procedures. Change from baseline to Week 12 will be recorded.
Change in Total Body Water | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Total body water will be assessed via TANITA BC-545N. Device output will be reported as percentage (%) or liters (L), depending on the measurement format. Changes from baseline to Week 12 will be evaluated.
Change in Depression Symptoms (Beck Depression Inventory) | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  Depressive symptoms will be evaluated using the Beck Depression Inventory (BDI).
Change in PCOS-Specific Quality of Life (PCOSQ-50) | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  The PCOSQ-50 questionnaire assesses PCOS-specific quality of life across multiple domains.
Change in Health-Related Quality of Life (SF-36) | Participants follow the dietrary intervention and are assessed at baseline and at the end of the 12-week intervention.
  The SF-36 evaluates general health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University Kurupelit Campus, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No